CLINICAL TRIAL: NCT03215992
Title: Diffuse Optical Tomography in Prostate Cancer Detection and Risk Stratification A Pilot Study
Brief Title: Optical Tomography in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Emerson Lim, Assistant Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAAL3709
Record Dates: First submitted 2017-07-04; First posted 2017-07-12 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Diffuse Optical Tomography
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Men diagnosed with prostate cancer (Other): This group will include men over the age of 18 suspected of having prostate cancer who will undergo an ultrasound guided transrectal prostate biopsy. Each study participant will undergo a standard prostate biopsy and DOT imaging using the Diffuse Optical Tomography (DOT) System will be performed at the same time.
  Interventions: Device: Diffuse Optical Tomography (DOT) System
- Men without prostate cancer (Other): This group will include men who do not have prostate cancer. Each study participant will undergo a standard prostate biopsy and DOT imaging using the Diffuse Optical Tomography (DOT) System will be performed at the same time.
  Interventions: Device: Diffuse Optical Tomography (DOT) System

INTERVENTIONS:
Device: Diffuse Optical Tomography (DOT) System — Diffuse optical tomography (DOT) is a novel imaging modality that uses low-intensity, near-infrared light to characterize tissue. As light of a specific wavelength travels through tissue, it is absorbed and scattered by different chromophores and cellular structures. Using four wavelengths of light allows the detection of four chromophores: oxyhemoglobin, deoxyhemoglobin, water and fat.

SUMMARY:
This study is looking to see if a new device, diffuse optical tomography (DOT), can detect prostate cancer. The investigators will also see if DOT can tell the difference between high risk and low risk prostate cancers.

DETAILED DESCRIPTION:
While some of these tools have helped to guide therapy in patients with prostate cancer, they are imperfect and as a result many men undergo unnecessary treatment for a disease that would not have caused their deaths. An improved method to risk stratify men with prostate cancer prior to definitive therapy may reduce the over-treatment rate, while maintaining or improving mortality.

Diffuse optical tomography (DOT) is a novel imaging modality that uses low-intensity, near-infrared light to characterize tissue. DOT analyzes the light being reflected and transmitted through tissue to generate three-dimensional images of chromophores and light scattering. As such, DOT serves as a functional imaging modality, measuring both tissue vascularity and architecture. The investigators believe that DOT will be able to detect prostate cancer in men suspected of the disease and will also be able to risk-stratify patients found to have prostate cancer to help guide treatment options. DOT may be able to directly measure two factors important in the prognosis of patients with prostate cancer: the Gleason score and microvessel density (MVD).

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years of age or older scheduled for transrectal prostate biopsy or radical prostatectomy at Columbia University Medical Center
* Signing consent for study imaging procedure and analysis of prostate biopsy

Exclusion criteria:

* Patients failing to meet the inclusion criteria
* Contraindication for magnetic resonance imaging

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Total number of subjects who are imaged using DOT and produce usable images | Up to 3 years
  Total number of subjects who produce usable images will be measured to assess feasibility of concurrent transrectal ultrasound guided (TRUS) biopsy/DOT imaging, which is defined as successfully imaging and generating usable DOT data in 60% of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Lim, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided